CLINICAL TRIAL: NCT01369628
Title: A Phase Ib, Multicenter, Open Label, Dose-Escalating, Repeat-Dose Trial to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Atacicept When Administered to Subjects With Lupus Nephritis on a Stable Regimen of Mycophenolate Mofetil (MMF) With or Without Corticosteroids
Brief Title: Atacicept in Lupus Nephritis Patients Taking Stable Regimen of Mycophenolate Mofetil
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Please see Purpose Statement below
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 700461_014
Record Dates: First submitted 2011-06-07; First posted 2011-06-09 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Lupus Nephritis
Keywords: Open label; Dose Escalating; Phase Ib
MeSH Terms: conditions — Lupus Nephritis | interventions — TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): 1 arm with the 3 following dose regimens:
  1. Regimen 1: Atacicept 25 mg weekly for 12 weeks
  2. Regimen 2: Atacicept 75 mg weekly for 12 weeks
  3. Regimen 3: Atacicept 150 mg weekly for 12 weeks
  Interventions: Drug: Atacicept

INTERVENTIONS:
Drug: Atacicept — 1. Regimen 1: Atacicept 25 mg weekly for 12 weeks
  2. Regimen 2: Atacicept 75 mg weekly for 12 weeks
  3. Regimen 3: Atacicept 150 mg weekly for 12 weeks

SUMMARY:
The sponsor electively terminated the study because the risk mitigation measures, deemed necessary after an unforeseen safety event, could not be effectively implemented within this protocol while maintaining study timelines within a reasonable time frame.

DETAILED DESCRIPTION:
This study will evaluate atacicept's effects in subjects who have lupus nephritis, at least 2 g/day of protein in the urine, and are already taking mycophenolate mofetil. The evaluations will include the concentrations of atacicept in the blood, the effects of atacicept on immunoglobulins (antibodies), and any side effects. The first subjects will be given a low dose. Following periodic reviews of the trial data, subsequent subjects are planned to receive one of 2 progressively higher doses of atacicept.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, ≥ 18 years of age, who provide written informed consent
* Subjects must have a diagnosis of SLE satisfying ≥ 4 of 11 ACR criteria, and must have had a renal biopsy during screening or within the previous 18 months demonstrating class III (A or A/C), IV (A or A/C), V, or concomitant III/V or IV/V LN as defined by the International Society of Nephrology/Renal Pathology Society (ISN/RPS).
* Subjects must have a urine protein: creatinine ratio ≥ 2 mg/mg (≥ 226.2 mg/mmol), and either a positive test for antinuclear antibody (ANA) (HEp-2 ANA ≥ 1:80) and/or anti-double stranded deoxyribonucleic acid (dsDNA) (≥ 30 IU/mL) at screening.
* Subjects must have started induction therapy for LN at least 5 months prior to Trial Day 1, be considered to have received continuous treatment for LN during the 5 months prior to Trial Day 1, and have received a stable dose of MMF ≥ 1 g/day, with or without corticosteroids, for at least 8 weeks prior to Trial Day 1.

Exclusion Criteria:

* Recent changes in immunosuppressant, ACD inhibitors for ARBs
* Use of azathioprine, cyclosporine, tacrolimus, or cyclophosphamide or other biologics within 8 weeks prior to Trial Day 1.
* Serum IgG < 6 g/L
* Estimated Glomerular Filtration Rate (GFR) ≤ 30 mL/min per 1.73 m2
* History of Demyelinating Disease
* Significant Hematuria and/or Proteinuria due to a reason(s) other than LN. Evaluation should be done according to the local standard of care
* Breast feed or pregnancy
* Legal Incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The nature (preferred terms) and incidence of AEs | 12 weeks
  Frequency tables summarizing the observed number of AEs by System Organ Class (SOC) and preferred term will be presented per regimen.
Proportion of subjects fulfilling criteria for an Atacicept dose modification due to an IgG decrease | 12 weeks
  Percentages of subjects fulfilling the criteria (prespecified in the protocol) for an atacicept dose modification due to a decrease in IgG will be presented.
The frequency and severity of laboratory abnormalities | 12 weeks
  The incidence of subjects given each atacicept regimen who have shifts from Baseline in serum creatinine, serum albumin, urinary protein, or Hematology test (counts of white blood cells, neutrophils, lymphocytes, platelets) of at least 2 grades will be presented. Grading will be classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 toxicity grading, using the worst grade post-baseline during the 12-week treatment period.

SECONDARY OUTCOMES:
The nature (preferred terms) and incidence of AEs | 36 weeks
  Frequency tables summarizing the observed number of AEs by System Organ Class (SOC) and preferred term will be presented per regimen.
Proportion of subjects fulfilling criteria for an Atacicept dose modification due to an IgG decrease | 36 weeks
  Percentages of subjects fulfilling the criteria (prespecified in the protocol) for an atacicept dose modification due to a decrease in IgG will be presented.
The frequency and severity of laboratory abnormalities | 36 weeks
  The incidence of subjects given each atacicept regimen who have shifts from Baseline in serum creatinine, serum albumin, urinary protein, or Hematology test (counts of white blood cells, neutrophils, lymphocytes, platelets) of at least 2 grades will be presented. Grading will be classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 toxicity grading, using the worst grade post-baseline during the 12-week treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- EMD Serono Inc., One Technology Place, Rockland, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/20302641
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/19743503
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/19395457
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/18050206
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/10801128